CLINICAL TRIAL: NCT05185544
Title: Combining Genomics and Imageomics to Predict the Sensitivity of Neoadjuvant Pemetrexed and Cisplatin Chemotherapy in Patients With Lung Adenocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2021-Zhan
Record Dates: First submitted 2021-12-18; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Sensitivity
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- neoadjuvant pemetrexed and cisplatin chemotherapy in patients with lung adenocarcinoma: neoadjuvant pemetrexed and cisplatin chemotherapy in patients with lung adenocarcinoma
  Interventions: Other: Neoadjuvant pemetrexed and cisplatin chemotherapy

INTERVENTIONS:
Other: Neoadjuvant pemetrexed and cisplatin chemotherapy — neoadjuvant pemetrexed and cisplatin chemotherapy in patients with lung adenocarcinoma

SUMMARY:
Combining genomics and imageomics to predict the sensitivity of neoadjuvant pemetrexed and cisplatin chemotherapy in patients with lung adenocarcinoma

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged between 18 and 75 years;
* 2. Lung adenocarcinoma;
* 3. The patient is able to receive neoadjuvant pemetrexed and cisplatin chemotherapy
* 4 .The patient is able to understand and comply with the study and has provided written informed consent.

Exclusion Criteria:

* 1. Patients with a history of lung surgery;
* 2. Postoperative pathology showed non-primary lung cancer;
* 3. Patients with a history of other tumors;
* 4. Patients with severe complications (coronary heart disease, valvular heart disease, end-stage renal disease, severe liver cirrhosis);
* 5. Unable to cooperate with the researchers because of dementia or cognitive decline
* 6. Other situations that are not in conformity with the standards and requirements of this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neoadjuvant pemetrexed and cisplatin chemotherapy in patients with lung adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor Regression Grade | 1-2 Weeks after enrollment (after Surgery)